CLINICAL TRIAL: NCT01713686
Title: Prospective, Multi-center, Pivotal Trial Evaluating the Safety and Effectiveness of the Ulthera® System for Improvement in Lines and Wrinkles of the Décolletage
Brief Title: Evaluation of the Ulthera System for the Treatment of the Decolletage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-129
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Chest Wrinkles
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Micro-focused Ultrasound with Visualization (MFU-V)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ulthera System Treatment (Experimental): A single triple-depth Ulthera System treatment of the decolletage delivering treatment at 4.5mm, 3.0mm and 1.5mm depths.
  Interventions: Device: Ulthera System Treatment

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™

SUMMARY:
This is prospective, multi-center clinical trial. Enrolled subjects will receive one Ulthera® treatment on the decolletage. Follow-up visits will occur at 90 and 180 days following treatment. Study images will be obtained pre-treatment, immediately post-treatment, and at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 35 to 70 years.
* Subject in good health.
* Moderate to severe skin lines and wrinkles on the décolletage; grade of ≥4 on a chest wrinkle scale.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating.
* Absence of physical conditions unacceptable to the investigator.
* Willingness and ability to provide written consent for study-required photography.
* Willingness and ability to provide written informed consent.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Scarring in areas to be treated.
* Tattoos in the areas to be treated.
* Patients with ports or defibrillators.
* Any open wounds or lesions in the area.
* Active and severe inflammatory acne in the region to be treated.
* Patients who have a history with keloid formation or hypertrophic scarring.
* Inability to understand the protocol or to give informed consent.
* Retinoid, microdermabrasion, or prescription level glycolic acid treatments to the décolletage area within two weeks prior to study participation or during the study.
* Marked décolletage asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin.
* History of chronic drug or alcohol abuse.
* History of autoimmune disease.
* Concurrent therapy that would interfere with the evaluation of the safety or effectiveness of the study device.
* Subjects who anticipate the need for surgery or overnight hospitalization during the study.
* Subjects who have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
* Concurrent enrollment in any study involving the use of investigational devices or drugs.
* Current smoker or history of smoking in the last one year.
* History of using the following prescription medications:

  1. Topical Retinoids to the area within the past two weeks;
  2. Antiplatelet agents/anticoagulants (Coumadin, Heparin, Plavix).
  3. Psychiatric drugs that would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc.
Locations (4):
- United States (4):
  - Laser Skin and Surgery Center of Northern California, Sacramento, California
  - Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc., San Diego, California
  - Denova Research, Chicago, Illinois
  - Tennessee Research Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Ulthera System Treatment: A single triple-depth Ulthera System treatment of the décolletage delivering treatment at 4.5mm, 3.0mm and 1.5mm depths.
  Ulthera System Treatment: Focused ultrasound energy delivered below the surface of the skin
Period: Overall Study
Arm/Group | Ulthera System Treatment
Started | 125 (129 enrolled, 125 treated. 2 withdrew consent prior to treatment; 2 excluded after enrollment.)
Completed | 110
Not Completed | 15
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Ulthera System Treatment
Number analyzed (Participants) | 125
Age, Continuous [Mean (Full Range); unit: years] | 56.7 [37.5 to 70.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 117
  Hispanic/Latino | 7
  Other | 1
Fitzpatrick's Sun-Reactive Skin Type [Number; unit: participants] — A classification for skin color:
  * Type I Pale white; blond or red hair; blue eyes; freckles - Always burns, never tans;
  * Type II White; fair; blond or red hair; blue, green or hazel eyes - Usually burns, tans minimally;
  * Type III Cream white; fair with any hair or eye color; quite common - Sometimes mild burn, tans uniformly;
  * Type IV Moderate brown; typical Mediterranean skin tone - Rarely burns, always tans well;
  * Type V Dark brown; Middle Eastern skin types - Very rarely burns, tans very easily;
  * Type VI Deeply pigmented dark brown to black - Never burns, tans very easily.
  participants
    Type I | 1
    Type II | 60
    Type III | 52
    Type IV | 12
    Type V | 0
    Type VI | 0
BMI [Mean (Full Range); unit: kg/m^2] | 24.7 [18.3 to 38.3]
Fabi/Bolton Score [Number; unit: participants] — 5-point photonumeric scale, with the following descriptors:
  1. Wrinkles absent
  2. Shallow lines, but visible
  3. Moderately deep lines
  4. Deep with well-defined lines
  5. Very deep with redundant folds
  participants
    Fabi/Bolton Score 1 | 0
    Fabi/Bolton Score 2 | 0
    Fabi/Bolton Score 3 | 0
    Fabi/Bolton Score 4 | 111
    Fabi/Bolton Score 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Reduction in Chest Wrinkles at 90 Days Post Treatment
Description: Assessment of improvement, in a blinded fashion, using a Chest Wrinkle Scale at 90 days post-treatment. However, during conduct of the trial, the Chest Wrinkle scale was deemed inadequate as a primary endpoint in this study. Therefore, conduct of a traditional blinded masked assessment, the gold-standard measure in aesthetics, was used as the primary endpoint,i.e., improvement in wrinkles and lines of the décolletage as determined by a blinded, masked, qualitative assessment of photographs at 90 days post-treatment compared to baseline.
  "Improvement" = a blinded evaluator assessed an "Improvement" when evaluating a masked, paired photo set and correctly chose the Post treatment photo.
  "Incorrect" = a blinded evaluator assessed an "Improvement" when evaluating a masked, paired photo set but incorrectly chose the Post treatment photo.
Time Frame: 90 Days post-treatment
Population: The analysis population was based on data from subjects completing a 90 day follow-up visit. Of the 116 subjects who returned for the D90 follow-up, 113 subjects had evaluable photographs. These photos were treated as 'missing' by the statistician and were not included in the denominator for the masked assessment analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Ulthera System Treatment
Number analyzed (Participants) | 113
percentage of participants
  Improvement | 69.9
  No change | 15.9
  Incorrect | 14.2

2. Secondary Outcome: Overall Aesthetic Improvement at 90 Days Post-treatment
Description: The overall level of aesthetic improvement at 90 Days post treatment compared to baseline was assessed using a Clinician Global Aesthetic Improvement Scale (CGAIS). The CGAIS is a 5-point scale with the following descriptors:
  1. Very much improved
  2. Much improved
  3. Improved
  4. No change
  5. Worse
  The scale was completed in two steps:
  * Based on a live assessment of the subject while referring to the subject's pre-treatment photographs; and
  * Based on a comparison of the subject's pre-treatment photographs to current post-treatment photographs.
  "Improved" = Very Much Improved + Much Improved + Improved
Time Frame: 90 days post-treatment
Population: This secondary outcome measure was based on 116 subjects completing a 90 day post-treatment visit.
Measure: Number; unit: percentage of participants
Arm/Group | Ulthera System Treatment
Number analyzed (Participants) | 116
percentage of participants
  Improved | 75.1
  No change | 24.1
  Worse | 0.9

3. Secondary Outcome: Overall Aesthetic Improvement at 180 Days Post-treatment
Description: The overall level of aesthetic improvement at 180 Days post treatment compared to baseline was assessed using a Clinician Global Aesthetic Improvement Scale (CGAIS). The CGAIS is a 5-point scale with the following descriptors:
  1. Very much improved
  2. Much improved
  3. Improved
  4. No change
  5. Worse
  The scale was completed in two steps:
  * Based on a live assessment of the subject while referring to the subject's pre-treatment photographs; and
  * Based on a comparison of the subject's pre-treatment photographs to current post-treatment photographs.
  "Improved" = Very Much Improved + Much Improved + Improved
Time Frame: 180 days post-treatment
Population: Analysis population was based the number of subjects completing a 180 day follow-up visit.
Measure: Number; unit: percentage of participants
Arm/Group | Ulthera System Treatment
Number analyzed (Participants) | 110
percentage of participants
  Improved | 66.4
  No Change | 30.0
  Worse | 3.6

4. Primary Outcome: Percentage of Participants With a Reduction in Chest Wrinkles at 180 Days Post Treatment
Description: Assessment of improvement, in a blinded fashion, using a Chest Wrinkle Scale at 180 days post-treatment. However, during conduct of the trial, the Chest Wrinkle scale was deemed inadequate as a primary endpoint in this study. Therefore, conduct of a traditional blinded masked assessment, the gold-standard measure in aesthetics, was used as the primary endpoint, improvement in wrinkles and lines of the décolletage as determined by a blinded, masked, qualitative assessment of photographs at 180 days .post-treatment compared to baseline.
  "Improvement" = a blinded evaluator assessed an "Improvement" when evaluating a masked, paired photo set and correctly chose the Post treatment photo.
  "Incorrect" = a blinded evaluator assessed an "Improvement" when evaluating a masked, paired photo set but incorrectly chose the Post treatment photo.
Time Frame: 180 days post treatment
Population: The analysis population was based on the Last Value Carried Forward (LVCF) analysis method for determining overall efficacy, i.e., if a D90 but not D180 value was present, the LVCF is the D90 value. Following this method, the analysis popullation was based on 116 subjects.
Measure: Number; unit: percentage of participants
Arm/Group | Ulthera System Treatment
Number analyzed (Participants) | 116
percentage of participants
  Improved | 66.4
  No Change | 11.2
  Incorrect | 22.4

5. Secondary Outcome: Subject Satisfaction at 90 Days Post-treatment
Description: Subject satisfaction was measured at 90 days post-treatment using a Patient Satisfaction Questionnaire (PSQ). A 5-point PSQ scale was used with the following descriptors:
  1. Very Satisfied
  2. Satisfied
  3. Neither Satisfied or Dissatisfied
  4. Dissatisfied
  5. Very Dissatisfied
  "Satisfied"= Very Satisfied + Satisfied
  "Dissatisfied"=Dissatisfied + Very Dissatisfied
Time Frame: 90 days post-treatment
Population: This secondary outcome measure was based on the responses provided from 116 subjects completing a 90 day post-treatment visit.
Measure: Number; unit: percentage of participants
Arm/Group | Ulthera System Treatment
Number analyzed (Participants) | 116
percentage of participants
  Satisfied | 65.5
  Neither Satisfied or Dissatisfied | 29.3
  Dissatisfied | 5.2

6. Secondary Outcome: Subject Satisfaction at 180 Days Post-treatment
Description: Subject satisfaction was measured at 180 days post-treatment using a Patient Satisfaction Questionnaire (PSQ). A 5-point PSQ scale was used with the following descriptors:
  1. Very Satisfied
  2. Satisfied
  3. Neither Satisfied or Dissatisfied
  4. Dissatisfied
  5. Very Dissatisfied
  "Satisfied" = Very Satisfied + Satisfied
  "Dissatisfied" = Dissatisfied + Very Dissatisfied
Time Frame: 180 days post-treatment
Population: This secondary outcome measure was based on the responses provided from 116 subjects completing a 180 day post-treatment visit.
Measure: Number; unit: percentage of participants
Arm/Group | Ulthera System Treatment
Number analyzed (Participants) | 110
percentage of participants
  Satisfied (satisfied and very satisfied) | 62.7
  Neither Satisfied nor Dissatisfied | 22.7
  Dissatisfied (dissatisfied and very dissatisfied) | 14.5

ADVERSE EVENTS:
Time Frame: Adverse events were followed for up to 6 months post-treatment or until event resolution.
Groups:
- Ulthera System Treatment: A single triple depth Ulthera System treatment of the décolletage delivering treatment at 4.5mm, 3.0mm and 1.5mm depths.
  Ulthera System Treatment: Focused ultrasound energy delivered below the surface of the skin
Arm/Group | Ulthera System Treatment
Serious Adverse Events (participants affected / at risk) | 0/125
Other Adverse Events (participants affected / at risk) | 83/125
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ulthera System Treatment (N=125)
Tenderness (Skin and subcutaneous tissue disorders) | 45 (45)
Bruising (Skin and subcutaneous tissue disorders) | 22 (22)
Pruitus (Skin and subcutaneous tissue disorders) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No